CLINICAL TRIAL: NCT00875407
Title: Feasibility of 123I-IBZM Scintigraphy (a D2 Agonist) in Patients With Pheochromocytoma (PHEO) and/or Paraganglioma (PGL) : Study Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008/09; 2008-A007932-52
Record Dates: First submitted 2009-04-01; First posted 2009-04-03 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Chromaffin-tissue Derived Tumors
MeSH Terms: interventions — 3-iodo-2-hydroxy-6-methoxy-N-((1-ethyl-2-pyrrolidinyl)methyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Scintigraphy in 123I-IBZM

SUMMARY:
Context. Nuclear imaging plays a central role in management of chromaffin-tissue derived tumors because tumor cells exhibit peptide receptors and proteins involved in metabolism that can be targeted with specific radiopharmaceutics. Recently, over expression dopamine-receptor D2 isoforms has been found in endocrine tumors.

Objective. The aim of the present study is to evaluate the feasibility of 123I-IBZM (a D2 agonist radiolabelled with 123I) in patients with PHEO and/or PGL. Diagnostic accuracy will be also compared to traditional SPECT imaging procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age + 18 years. The women in ages to procreate have to have an effective contraception or a negative pregnancy test (in the absence of effective contraception) Having a radiological and functional imaging (balance sheet(assessment) pré--IBZM) considered adapted and complete for the pathology.
* Having a phéochromocytome or a paragangliome proving a surgical operation in view of the data of the balance sheet(assessment) pré--IBZM.
* With or without allergy in the iodine.

Exclusion Criteria:

* NEM2A or 2B.
* Malignant Forms which do not recover from an even partial, surgical gesture(movement).
* Pregnant Women or in the course of feeding.
* Women in age to procreate without effective contraception, with positive pregnancy test.
* Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The aim of the present study is to evaluate the feasibility of 123I-IBZM (a D2 agonist radiolabelled with 123I) in patients with PHEO and/or PGL. Diagnostic accuracy will be also compared to traditional SPECT imaging procedures. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: DAVID TAIEB, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique-Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Saveanu A, Sebag F, Guillet B, Archange C, Essamet W, Barlier A, Palazzo FF, Taieb D. Targeting dopamine receptors subtype 2 (D2DR) in pheochromocytomas: head-to-head comparison between in vitro and in vivo findings. J Clin Endocrinol Metab. 2013 Dec;98(12):E1951-5. doi: 10.1210/jc.2013-2269. Epub 2013 Sep 5. PMID 24009136